CLINICAL TRIAL: NCT02642432
Title: A Single Arm, Open-label Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 1, 2, 4, 5 or 6 Infection and Compensated Cirrhosis (EXPEDITION-1)
Brief Title: A Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 1, 2, 4, 5 or 6 Infection and Compensated Cirrhosis
Acronym: EXPEDITION-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-172; 2015-003797-32 (EudraCT Number)
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Virus Infection; Chronic Hepatitis C; Compensated Cirrhosis
Keywords: HCV Genotype 1; HCV Genotype 4; HCV Genotype 2; Cirrhotic; Interferon-Free; Compensated Cirrhosis; HCV Genotype 5; Hepatitis C; HCV Genotype 6
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-493/ABT-530 (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET

SUMMARY:
The purpose of this study is to assess the safety and efficacy of ABT-493/ABT-530 following 12 weeks of treatment in adults with chronic Hepatitis C Virus Infection genotype 1, 2, 4, 5 or 6 infection and compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Screening laboratory result indicating hepatitis C virus (HCV) Genotype 1, 2, 4, 5 or 6 (GT1,2,4,5,6) infection
* Chronic HCV infection
* Subject must be HCV treatment-naïve or have failed prior HCV treatment
* Subject must have documented compensated cirrhosis and no current or past clinical evidence of decompensated liver disease

Exclusion Criteria:

* Positive test result at screening for Hepatitis B surface antigen or anti-human immunodeficiency virus (anti-HIV) antibody
* HCV genotype performed during screening indicating co-infection with more than 1 HCV genotype
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-493/ABT-530

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Background] Forns X, Lee SS, Valdes J, Lens S, Ghalib R, Aguilar H, Felizarta F, Hassanein T, Hinrichsen H, Rincon D, Morillas R, Zeuzem S, Horsmans Y, Nelson DR, Yu Y, Krishnan P, Lin CW, Kort JJ, Mensa FJ. Glecaprevir plus pibrentasvir for chronic hepatitis C virus genotype 1, 2, 4, 5, or 6 infection in adults with compensated cirrhosis (EXPEDITION-1): a single-arm, open-label, multicentre phase 3 trial. Lancet Infect Dis. 2017 Oct;17(10):1062-1068. doi: 10.1016/S1473-3099(17)30496-6. Epub 2017 Aug 14. PMID 28818546
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 35-day screening period.
Period: Overall Study
Arm/Group | ABT-493/ABT-530
Started | 146
Completed | 138
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Withdrew Consent | 1
Not completed — Lost to Follow-up | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.12 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 146
percentage of participants | 99.3 [98.0 to 100.0]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Treatment Weeks 1, 2, 4, 8, and 12 (end of treatment) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 146
percentage of participants | 0.0 [0.0 to 2.6]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 144
percentage of participants | 0.7 [0.1 to 3.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE event with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ABT-493/ABT-530
Serious Adverse Events (participants affected / at risk) | 11/146
Other Adverse Events (participants affected / at risk) | 63/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 (N=146)
GASTRIC ULCER (Gastrointestinal disorders) | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1
ENDOPHTHALMITIS (Infections and infestations) | 1
RECTAL ABSCESS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
TUMOUR MARKER INCREASED (Investigations) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
SYNCOPE (Nervous system disorders) | 1
ALCOHOL ABUSE (Psychiatric disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 (N=146)
DIARRHOEA (Gastrointestinal disorders) | 12
NAUSEA (Gastrointestinal disorders) | 13
FATIGUE (General disorders) | 27
URINARY TRACT INFECTION (Infections and infestations) | 9
HEADACHE (Nervous system disorders) | 20
PRURITUS (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.